CLINICAL TRIAL: NCT00095901
Title: A Phase II Study Of Capecitabine In Previously Treated, Recurrent And/Or Metastatic Nasopharyngeal Carcinoma
Brief Title: Capecitabine For Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Wirth, Lori MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-384; P30CA006516 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Capecitabine (Xeloda 4:14. ) 150 mg and 500 mg tablets. Capecitabine will be administered at a dose of 1000 mg/m2 twice daily, for a total daily dose of 2000 mg/m 2. Capecitabine will administered P.O. or per G-tube B.I.D. for 14 days, followed by a one-week rest period in 3-week cycles.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This study plans to examine the effects of Capecitabine administered as an oral chemotherapy drug in participants with nasopharyngeal cancer.

Capecitabine is an oral prodrug. A "prodrug" is a drug that is converted within the body into its active form that has medical effects. Capecitabine is a prodrug of 5-fluorouracil (5-FU), which is a chemotherapy agent frequently used to treat head and neck cancers. Capecitabine is absorbed through the gastrointestinal tract and is converted to 5-FU. Capecitabine (Xeloda9) has been tested in subjects with colorectal and breast cancers, and shown to be effective in those cancers. Likewise, 5-FU has shown benefit when administered as a continuous infusion for those with nasopharyngeal cancers. Since Capecitabine is a prodrug of 5-FU, it is possible that similar results will be achieved.

RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have locally recurrent or metastatic nasopharyngeal cancer.

DETAILED DESCRIPTION:
This is a nonrandomized, multicenter study.

- Patients receive oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days.

ELIGIBILITY:
* Inclusion Criteria

  * To be eligible for inclusion, each patient must fulfill each of the following criteria:
  * Provide written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
  * At least 18 years of age.
  * Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (see Appendix C).
  * Histologically confirmed nasopharyngeal carcinoma, WHO types I, II or III, with recurrent locoregional and/or metastatic disease. Primary cancers of the nasal cavity or paranasal sinuses, sinonasal neuroendocrine carcinomas or primary malignancies of the salivary gland will NOT be eligible.
  * Have received at least one, but no more than 2, prior chemotherapy regimens for recurrent and/or metastatic disease. Patients with recurrent locoregional and/or metastatic NPC who are unable to tolerate a platinum-based chemotherapy due to previous treatment with a platinum or a condition that precludes their use will also be eligible.
  * Have tumor tissue available for EBER analysis, if not already done.
  * Have at least one measurable lesion according to the RECIST criteria (see Appendix B) which has not been irradiated within 6 months of enrollment. Pleural effusion and bone metastases are not considered measurable. Minimum indicator lesion size: ≥ 10 mm measured by spiral CT or ≥ 20 mm measured by conventional techniques.
  * Have a negative serum or urine pregnancy test within 7 days prior to registration in female patients of childbearing potential.
* Exclusion Criteria

  * Patients who fulfill any of the following criteria will be excluded:
  * Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Women or men of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
  * Life expectancy <3 months.
  * Serious, uncontrolled, concurrent infection(s).
  * Prior fluoropyrimidine therapy within 6 months of enrollment. Subjects with previous 5-FU or other fluoropyrimidine treatment are eligible, if ≥ 6 months has elapsed since this previous therapy.
  * Prior unanticipated severe reaction to fluoropyrimidine therapy, or known extreme sensitivity to 5-FU.
  * Completion of previous chemotherapy regimen < 4 weeks prior to the start of study treatment, or with related toxicities unresolved prior to the start of study treatment.
  * Previous radiotherapy < 4 weeks prior to the start of study treatment.
  * Other malignancy within the last five years, except non-melanoma skin and in-situ cervical cancer.
  * Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
  * Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
  * Evidence of central nervous system (CNS) metastases (unless CNS metastases have been stable for > 3 months) or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
  * Major surgery within 4 weeks of the start of study treatment, without complete recovery.
  * Malabsorption syndrome of the upper gastrointestinal tract.
  * Any of the following laboratory values:

    * Abnormal hematologic values (neutrophils < 1.5 x 10 9/L, platelet count < 100 x 10 9/L)
    * Impaired renal function (estimated creatinine clearance <30 ml/min as calculated with Cockroft-Gault equation or serum creatinine > 1.5 x upper normal limit).
    * Note: In patients with moderate renal impairment (estimated creatinine clearance 30-50 mL/min) at baseline, a dose reduction to 75% of the capecitabine starting dose is recommended.
    * Serum bilirubin > 1.5 x upper normal limit.
    * ALT, AST > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
    * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease).
  * Unwillingness to give written informed consent.
  * Unwillingness to participate or inability to comply with the protocol for the duration of the study.
  * Other serious uncontrolled medical conditions that the investigator feels might compromise study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Rate of Response | 4 weeks
  Tumor response rate based on tumor measurement (according to the nasT criteria). Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Correlation of Epstein-Barr virus (EBV) with response as assessed by a two-sample t-test with arcsin approximation | Baseline and every 2 cycles
Correlation of EBV status to thymidine phosphorylase expression as assessed by Fischer's exact test | Basleine and every 2 cycles
Correlation of response to thymidine phosphorylase expression as assessed by Fischer's exact test | Baseline and every 2 cycles
Rate of Progression Free Survival | Study Day 1 to the date of first known disease progression, or the date of death if the patient
Rate of Overall Survival | Study Day 1 to the date of death or the last date patient was known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Wirth, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No